CLINICAL TRIAL: NCT04767269
Title: Efficacy of Cuminum Cyminum Herbal Preparation in Inhibition of Plaque and Gingivitis
Brief Title: Efficacy of Cuminum Cyminum Herbal =Preparation in Inhibition of Plaque and Gingivitis.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, DR SURINDER SACHDEVA, Professor, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MaharishiMu2012
Record Dates: First submitted 2021-02-09; First posted 2021-02-23 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Chronic Gingivitis
Keywords: Mouthwash; chlorhexidine; stain

STUDY DESIGN:
Intervention Model Description: 1. Group phase A
  2. Group phase B
  3. Group phase C
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cuminum cyminum mouthwash (Experimental): cuminum cyminum mouthwash in chronic gingivitis patients
  Interventions: Drug: Cuminum Cyminum
- herbal mouthwash (Active Comparator): herbal mouthwash in chronic gingivitis patients
  Interventions: Drug: herbal Mouthwash

INTERVENTIONS:
Drug: Cuminum Cyminum — Cuminum Cyminum mouthwash in chronic gingivitis patients
  Other Names: Cuminum Cyminum mouthwash
  Arms: cuminum cyminum mouthwash
Drug: herbal Mouthwash — herbal mouthwash in chronic gingivitis patients
  Other Names: herbal mouthwash in chronic gingivitis patients
  Arms: herbal mouthwash

SUMMARY:
Present work was to investigate the possible efficacy of 0.2% cuminum cyminum herbal preparation as an antiplaque and antigingivitis agent when compared with chlorhexidine.

DETAILED DESCRIPTION:
To evaluate and compare the efficacy of 0.2% cuminum cyminum herbal preparation against 0.2% chlorhexidine by various clinical parameters i.e. plaque index, gingival index and sulcus bleeding index.

ELIGIBILITY:
Inclusion Criteria:

* volunteers with minimum 20 natural teeth without restoration.
* cooperative
* motivated and committed to participate in the trial period.

Exclusion Criteria:

* Antibiotic or anti-inflammatory therapy in previous month.
* Any known allergy/ hypersensitivity to any product used in trial.

Ages: 23 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
PLAQUE INDEX | changes from baseline to 8 days
  PLAQUE INDEX: Turesky-Gilmore-Glickman Modification of Quigley Hein 1962
Gingival Index | changes from baseline to 8 days
  Gingival Index: Loe H ans Silness 1963
Bleeding on probing | changes from baseline to 8 days
  Bleeding on probing: Muhlemann HR and Son 1971

CONTACTS AND LOCATIONS:
Overall Officials: surinder sachdeva, M.D.S., Principal Investigator — PROFESSOR
Locations (1):
- Department of Periodontology, M.M. College of Dental Sciences and Research., Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Southern EN, McCombs GB, Tolle SL, Marinak K. The comparative effects of 0.12% chlorhexidine and herbal oral rinse on dental plaque-induced gingivitis. J Dent Hyg. 2006 Winter;80(1):12. Epub 2006 Jan 1. PMID 16451766
- [Background] Salgado AD, Maia JL, Pereira SL, de Lemos TL, Mota OM. Antiplaque and antigingivitis effects of a gel containing Punica granatum Linn extract: a double-blind clinical study in humans. J Appl Oral Sci. 2006 Jun;14(3):162-6. doi: 10.1590/s1678-77572006000300003. PMID 19089066
- [Background] Bettaieb I, Bourgou S, Wannes WA, Hamrouni I, Limam F, Marzouk B. Essential oils, phenolics, and antioxidant activities of different parts of cumin (Cuminum cyminum L.). J Agric Food Chem. 2010 Oct 13;58(19):10410-8. doi: 10.1021/jf102248j. PMID 20809647